CLINICAL TRIAL: NCT06156358
Title: Blood Indices as Predictors of Anastomotic Leak After Colorectal Surgery - Is It Useful? A Retrospective Analysis.
Brief Title: Indicators of Anastomotic Leak After Colorectal Surgery
Status: Completed | Type: Observational
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Dr. Mai Kadi, Assistant professor, King Abdulaziz University
Other Study IDs: AMSCRCL
Record Dates: First submitted 2023-11-26; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
We reviewed the patient underwent colorectal surgery with anastomosis and identified patients with anastomotic leak. Then we started to figure out what blood investigation could be related to anastomotic leak.

ELIGIBILITY:
Inclusion Criteria:

* Patient underwent colorectal surgery with anastomosis

Exclusion Criteria:

* Patient has no colon or rectum as part of anastomosis
* Patient with more than one procedure within 6 month

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients underwent abdominal surgery with colon or rectum anastomosis
Sampling Method: Non-Probability Sample
Enrollment: 441 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-07-03 (Actual)

PRIMARY OUTCOMES:
Accuracy of blood investigations in detecting anastomotic leak | JAN 2015 - DEC 2022

IPD SHARING:
Plan to Share IPD: Undecided
Data will provided upon reasonable request